CLINICAL TRIAL: NCT00815906
Title: An Ascending Single Dose Study Of The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of SBI-087 Administered To Japanese Subjects With Rheumatoid Arthritis
Brief Title: Study Evaluating Single Doses Of SBI-087 In Japanese Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Emergent Product Development Seattle LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3227K1-1001; B2261002
Record Dates: First submitted 2008-12-18; First posted 2008-12-31 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — SBI-087

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SBI-087 0.15 mg IV (Experimental)
  Interventions: Drug: SBI-087
- SBI-087 0.5 mg IV (Experimental)
  Interventions: Drug: SBI-087
- SBI-087 100 mg SC (Experimental)
  Interventions: Drug: SBI-087
- SBI-087 200 mg SC (Experimental)
  Interventions: Drug: SBI-087

INTERVENTIONS:
Drug: SBI-087 — IV, Single dose
  Arms: SBI-087 0.15 mg IV
Drug: SBI-087 — IV, Single dose
  Arms: SBI-087 0.5 mg IV
Drug: SBI-087 — SC, Single dose
  Arms: SBI-087 100 mg SC
Drug: SBI-087 — SC, Single dose
  Arms: SBI-087 200 mg SC

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single doses of SBI-087 in Japanese subjects with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Must meet American College of Rheumatology criteria for rheumatoid arthritis with functional class I to III.
* Rheumatoid arthritis disease onset at >16 years of age and duration of disease at least 6 months.
* Men or women of nonchildbearing potential (WONCBP), aged 20 to 70 years, inclusive at the screening visit.

Exclusion Criteria:

* Any significant health problems other than rheumatoid arthritis.
* Treatment of greater than 10 mg of prednisone per day.
* Therapy with immunosuppressants within 6 months before study day 1

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as determined by the number and severity of adverse events at the different dose levels | 12 months

SECONDARY OUTCOMES:
To describe the single-dose PK and PD profiles (B-cell count) after a SBI-087 administration in subjects with RA | 12 months
To evaluate the effect of a pretreatment regimen on the occurrence of systemic reactions following SC administration of 100 mg or 200 mg SBI-087 | 12 month
To investigate if changes in biomarkers (eg, complement activation markers, B-cells, CRP, IgE and tryptase levels) are related to the occurrence of systemic reactions on the day of infusion or injection of SBI-087 | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Japan (7):
  - Pfizer Investigational Site, Ehime
  - Pfizer Investigational Site, Fukui
  - Pfizer Investigational Site, Kanagawa
  - Pfizer Investigational Site, Miyagi
  - Pfizer Investigational Site, Ōita
  - Pfizer Investigational Site, Shizuoka
  - Pfizer Investigational Site, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3227K1-1001&StudyName=Study%20Evaluating%20Single%20Doses%20Of%20SBI-087%20In%20Japanese%20Subjects%20With%20Rheumatoid%20Arthritis